CLINICAL TRIAL: NCT03803709
Title: Dietary Fiber Intake in Alcohol-dependent Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 190616V1; 2017/04JUL/354 (Other: Ethics Committee CEHF)
Record Dates: First submitted 2018-12-13; First posted 2019-01-15 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2018-12

CONDITIONS: Alcoholism
Keywords: dietary fibers; alcohol-dependent
MeSH Terms: conditions — Alcoholism | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): * maltodextrin received at 4g/day on day 3 and 4
  * maltodextrin received at 8g/day from day 5 to 14
  * maltodextrin received at 16g/day from day 15 to 20
  Interventions: Dietary Supplement: placebo
- inulin (Experimental): * inulin received at 4g/day on day 3 and 4
  * inulin received at 8g/day from day 5 to 14
  * inulin received at 16g/day from day 15 to 20
  Interventions: Dietary Supplement: inulin

INTERVENTIONS:
Dietary Supplement: inulin — inulin given at different dosis from day 3 to day 20
  Arms: inulin
Dietary Supplement: placebo — maltodextrine given at different dosis from day 3 to day 20
  Arms: placebo

SUMMARY:
The alcohol problem affects 7.5% of the population in Europe and represents a major public health problem. Alcoholism is also a major cause of undernutrition. Diet is a major factor influencing the composition of the intestinal microbiota and previous studies, carried out at Saint-Luc clinics and catholic university of Louvain, show that alcoholic patients suffer from dysbiosis, that is a significant alteration of the gut microbiota. The investigator's preliminary studies, carried out at the Integrated Unit of Hepatology of Saint-Luc Clinics, have shown that alcohol represents more than 40% of total caloric intake in alcohol-dependent patients. In addition, alcoholic patients have an insufficient intake of dietary fiber, that is to say a contribution lower than the Belgian nutritional recommendations. Indeed, the Conseil Supérieur de la Santé recommends a total amount of dietary fiber equal to or greater than 25 grams per day to ensure correct intestinal function. Fructan-type dietary fiber (inulin and fructo-oligosaccharides) is found naturally in many fruits and vegetables (Jerusalem artichokes, asparagus, artichokes, onions, garlic, chicory roots, bananas). They are neither absorbed nor digested by human enzymes but fermented selectively by intestinal bacteria.

A good digestive tolerance to dietary fiber supplementation has been observed in healthy subjects as well as in obese patients, in previous studies conducted at catholic university of Louvain and Saint-Luc clinics. However, a nutritional rebalance via fiber supplementation and digestive fiber tolerance have never been tested in an alcohol-dependent population.

The primary objectives of this academic research project in nutrition, carried out in alcohol-dependent patients, are as follows:

1. restore a nutritional balance as recommended by the Conseil Supérieur de la Santé via a dietary fiber intake
2. to study digestive tolerance to fibers
3. to study the intestinal and psychological well-being related to a fiber intake

Depending on the results obtained during the achievement of the primary objectives, the biological samples (blood, stool) collected during the study will be used to analyze the composition of the intestinal microbiota and the plasma markers associated with intestinal function.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* aged between 18 and 65
* caucasian
* French speaking
* alcohol drunk less than 48h before day 1

Exclusion Criteria:

* another addiction, except smoking
* psychiatric comorbidity on axe 1 of Diagnostic and Statistical Manual-IV
* antibiotic, probiotic or fibers recent (<2 months) treatment (or other molecule modifying intestinal transit)
* Non-steroidial anti-inflammatory drug or glucocorticoids recently taken (<1 month)
* obesity: Body Mass Index<30
* bariatric surgery
* Type 1 or 2 diabetes
* chronic inflammatory diseases (Crohn disease, coeliac disease, rheumatoid arthritis)
* cirrhosis or Advanced hepatic fibrosis (Fibroscan > or = F3)
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-04 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in diet profile | on Day 2 and Day 19
  This tool is based on the one adapted to alcoholic patients at Saint Luc Hospital. It consists of two parts to allow cross-checking of data (redundancy) and to measure separate information:
  General: it is implemented a Food Frequency Questionnaire (FFQ) in order to investigate the general diet profile.
  Daily: it resumes the sequencing of a full day which allows to verify the information previously obtained as well as to precisely identify the moments of consumption of alcoholic and non-alcoholic inputs.
  This 7-day recall will be carried out at two times: week T1 for reminder of the week before hospitalization then T2 for reminder of the week back home. In this last case, this anamnesis will be done by interview, but also on the basis of the diary filled by the patient in T2, in order to optimize the accuracy of the data.

SECONDARY OUTCOMES:
Alimentary book | From day 1 to day 21
  The patient will have to fill in this book every day
Quantitative evaluation of intakes | on Day 2 and Day 19
  The meals will be weighted before and after eating
Alimentation history | On day 21
  This questionnaire makes it possible to further investigate the patient's diet before the episode of alcoholism in his adult and child life. The aim is to assess whether it is closer to a healthy diet (Mediterranean diet or dash diet) or a Western diet type. It is based on the recall technique and performed by a qualified dietician.
Change in mood | on Day 2 and Day 19
  Beck Depression Inventory (score 0-63). Higher score indicates higher depression level.
Change in anxiety | on Day 2 and Day 19
  State-Trait Anxiety Inventory (score 20-80). Higher score indicates higher anxiety level.
Change in alcohol craving | on Day 2 and Day 19
  Obsessive Compulsive Drinking Scale: a total score (= obsession + compulsion) (0-40) and 2 sub-scores (Obsession (0-20) and Compulsion (0-20)) are calculated. Higher score indicates higher craving level.
Change in impulsivity | on Day 2 and Day 19
  Urgency Premeditation Perseverance Sensation seeking impulsive behavior scale: score of different subscales are calculated: "urgency"(0-48), "lack of premeditation"(0-44), "lack of perseverance"(0-40), "sensation seeking"(0-48). Higher score in the different subscales indicates higher impulsivity level.
Change in selective attention | on Day 2 and Day 19
  William Lennox attention tests
Change in work memory | on Day 2 and Day 19
  Brown-Peterson's tasks
Change in flexibility | on Day 2 and Day 19
  Trail making test
Change in inhibition | on Day 2 and Day 19
  Scoop's tasks
Change in decision making | on Day 2 and Day 19
  Iowa gambling's task
Change in trauma | on Day 2 and Day 19
  Post-traumatic diagnostic scale: calculation of score is complex and described in the related publication Hearn, M, Ceschi, G., Brillon, P, Fürst, G., & Van der Linden, M. (2012). A French adaptation of the Post-traumatic Diagnostic scale. Canadian Journal of Behavioural Science, 44, 16-28.
Change in intestine integrity | on Day 2 and Day 19
  It will be determined by blood sample (LPS level)
Change in albumin, pre-albumin and zinc concentration | on Day 2 and Day 19
  It will be determined by blood sample
Change in intestinal permeability | on Day 2 and Day 19
  Patients will ingest 50microCurie of 51Chrome-Ethylenediamintetraacetic prepared in a Nutridrink®. This molecule is not normally absorbed by the intestine except when there is an increase in intestinal permeability (paracellular passage following rupture of tight junctions). The molecule is then filtered by the kidney and is found in the urine. A 24h urine collection will be carried out to measure the radioactivity emitted by 51Chrome-Ethylenediamintetraacetic
Change in fecal albumin concentration | on Day 2 and Day 19
  A stool sample will be collected to analyze a marker of intestinal permeability: fecal albumin
Intestinal permeability | On day 3
  a duodenal biopsy will be collected and the expression of the tight junctions regulating the intestinal permeability will be analyzed by sectional immunofluorescence and quantitative Polymerase Chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amadieu C, Ahmed H, Leclercq S, Koistinen V, Leyrolle Q, Starkel P, Bindels LB, Laye S, Neyrinck AM, Karkkainen O, De Timary P, Hanhineva K, Delzenne NM. Effect of inulin supplementation on fecal and blood metabolome in alcohol use disorder patients: A randomised, controlled dietary intervention. Clin Nutr ESPEN. 2025 Apr;66:361-371. doi: 10.1016/j.clnesp.2025.01.046. Epub 2025 Jan 27. PMID 39864520
- [Derived] Amadieu C, Maccioni L, Leclercq S, Neyrinck AM, Delzenne NM, de Timary P, Starkel P. Liver alterations are not improved by inulin supplementation in alcohol use disorder patients during alcohol withdrawal: A pilot randomized, double-blind, placebo-controlled study. EBioMedicine. 2022 Jun;80:104033. doi: 10.1016/j.ebiom.2022.104033. Epub 2022 Apr 28. PMID 35490461
- [Derived] Amadieu C, Coste V, Neyrinck AM, Thijssen V, Leyrolle Q, Bindels LB, Piessevaux H, Starkel P, de Timary P, Delzenne NM, Leclercq S. Restoring an adequate dietary fiber intake by inulin supplementation: a pilot study showing an impact on gut microbiota and sociability in alcohol use disorder patients. Gut Microbes. 2022 Jan-Dec;14(1):2007042. doi: 10.1080/19490976.2021.2007042. PMID 34923905
- [Derived] Amadieu C, Leclercq S, Coste V, Thijssen V, Neyrinck AM, Bindels LB, Cani PD, Piessevaux H, Starkel P, de Timary P, Delzenne NM. Dietary fiber deficiency as a component of malnutrition associated with psychological alterations in alcohol use disorder. Clin Nutr. 2021 May;40(5):2673-2682. doi: 10.1016/j.clnu.2021.03.029. Epub 2021 Mar 30. PMID 33933733